CLINICAL TRIAL: NCT00223821
Title: Enhancing Conservative Treatment for Urge Incontinence
Acronym: COMBO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2899-R
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Results first posted 2013-12-19 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2013-10

CONDITIONS: Urinary Incontinence
Keywords: Behavior Therapy; Behavioral Medicine; Behavioral Research; Behavioral Sciences; Combined Modality Therapy; Drug Therapy; Overactive bladder; Treatment Outcome; Urge incontinence; Urinary incontinence
MeSH Terms: conditions — Urinary Incontinence; Urinary Bladder, Overactive; Urinary Incontinence, Urge | interventions — oxybutynin; Tolterodine Tartrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Drug Therapy Aone (Active Comparator): Oxybutynin chloride, extended-release, individually-titrated
  Interventions: Drug: Oxybutynin chloride, extended-release, individually-titrated
- Drug Therapy + Behavioral Training (Experimental): Drug Therapy + Behavioral Training: Individually-titrated, extended-release oxybutynin chloride with management of side-effects. Behavioral training consists of teaching urge suppression strategies and pelvic floor muscle training.
  Interventions: Drug: Oxybutynin chloride, extended-release, individually-titrated; Behavioral: Behavior Training

INTERVENTIONS:
Drug: Oxybutynin chloride, extended-release, individually-titrated — Individually-titrated, extended-release oxybutynin chloride with management of side-effects.
  Other Names: Ditropan XL
Behavioral: Behavior Training — Behavioral training consists of teaching urge suppression strategies and pelvic floor muscle training.
  Arms: Drug Therapy + Behavioral Training

SUMMARY:
The primary objective of this project is to evaluate whether enhancing drug therapy with components of behavioral training, including pelvic floor muscle rehabilitation, results in better outcomes than drug therapy alone for urge incontinence in community-dwelling women.

DETAILED DESCRIPTION:
Urinary incontinence in women is a major problem with significant medical, psychological, and social consequences. Previous research on urge incontinence, a common form of incontinence, has demonstrated that behavioral and drug interventions are effective, but do not cure most patients. Thus there is a need to improve conservative treatment for urge incontinence in women. The primary objective of this project is to evaluate whether enhancing drug therapy with components of behavioral training, including pelvic floor muscle rehabilitation, results in better outcomes than drug therapy alone for urge incontinence in community-dwelling women. This project is a randomized controlled clinical trial. Sixty-four women with predominantly urge incontinence have been randomized. Stratification and blocked randomization procedures are used to assign a subject to 8 weeks of drug therapy alone or 8 weeks of drug therapy enhanced with components of behavioral training that can be administered in most any outpatient clinic. The drug therapy is extended release oxybutynin, a well-established pharmacologic agent with a state of the art drug delivery system that has the lowest rates of side-effect. The behavioral treatment is an innovative, comprehensive, behavioral training program, which includes pelvic floor muscle rehabilitation, teaching urge suppression and other skills to improve bladder control, and self-monitoring with bladder diaries. Bladder diaries completed by subjects before and after the treatment are used to calculate reduction in the frequency of incontinence. Secondary outcomes measures include a patient satisfaction questionnaire and three impact/quality of life measures (Incontinence Impact Questionnaire, Uro-Genital Distress Index, SF-12 Health Survey). The second objective of the study is to examine the cost-effectiveness of adding behavioral components to drug therapy. With the changing health care environment, there is increased concern with the costs of providing treatment. This project will compare the relative costs and value of combined intervention using the methods of cost-effectiveness analysis, the most widely adopted method for the economic evaluation of health interventions. The third objective of the study is to examine further the mechanisms by which these therapies reduce incontinence, including changes in bladder capacity, thresholds for bladder sensation, pelvic muscle strength, use of pelvic muscles in response to the sensation of urgency and frequency of urination. Pre-post changes in these parameters are measured to examine the effects of the treatment on these variables, and structural equation modeling will be used to examine whether changes in each of these measures are related to treatment outcome.

ELIGIBILITY:
Inclusion Criteria:

Participants in this study were ambulatory, community-dwelling women (veterans and nonveterans) with persistent urge or predominantly urge incontinence.

Participants must:

1. Be ambulatory.
2. Be able to come to the clinic for treatment.
3. Report urge incontinence.
4. Report incontinence occurring at least twice per week on average.
5. Report incontinence persisting for at least three months.
6. Not have received behavioral therapy in the University of Alabama at Birmingham (UAB) Continence Clinic or Department of Veterans Affairs (VA) Continence Clinic.
7. In the clinical interview, the subject must report involuntary loss of urine associated with a strong desire to void and that the condition has persisted for at least three months.
8. At least two urge accidents on the 7-day baseline bladder diary, and the number of urge accidents must exceed the number of other types of accidents.
9. On urodynamic evaluation, there must be cystometric evidence of bladder dysfunction, either: detrusor instability or maximal cystometric capacity is less than 400 ml.

Exclusion Criteria:

1. Continual leakage.
2. Urinary tract infection (defined as growth of greater than 10,000 colonies per ml of a urinary pathogen on urine culture).
3. Fecal impaction.
4. Uncontrolled metabolic problem.
5. Post-void residual volume > 150 ml.
6. Hematuria on microscopic examination in the absence of infection. A urologic consultation will be recommended and enrollment will depend on agreement between the urologist and geriatrician (co-PI) that entry into treatment protocol is not contraindicated.
7. Severe uterine prolapse (prolapse reaching the vaginal introitus).
8. Decompensated congestive heart failure, diagnosed by history or physical exam.
9. Impaired mental status. (<24 on Folstein's Mini-Mental State Exam).
10. Uncontrolled narrow angle glaucoma.
11. Gastric retention (by medical history).
12. Hypersensitivity to oxybutynin.
13. Current use of anticholinergic agents for detrusor instability. Subjects on these medications will be asked to discontinue them for the duration of the study. Evaluation will be delayed until the drug(s) have been discontinued for 2 weeks.
14. If on diuretic, dose stable for less than three months.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2003-09; Primary Completion 2008-11 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn L. Burgio, PhD MA BA, Principal Investigator — Birmingham, Alabama VA Medical Center
Locations (1):
- Birmingham VA Medical Center, Birmingham, Alabama, United States

REFERENCES:
- [Result] Burgio KL, Goode PS, Richter HE, Markland AD, Johnson TM 2nd, Redden DT. Combined behavioral and individualized drug therapy versus individualized drug therapy alone for urge urinary incontinence in women. J Urol. 2010 Aug;184(2):598-603. doi: 10.1016/j.juro.2010.03.141. Epub 2010 Jun 19. PMID 20639023
- [Derived] Funada S, Yoshioka T, Luo Y, Sato A, Akamatsu S, Watanabe N. Bladder training for treating overactive bladder in adults. Cochrane Database Syst Rev. 2023 Oct 9;10(10):CD013571. doi: 10.1002/14651858.CD013571.pub2. PMID 37811598

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were community-dwelling women with urge predominant incontinence recruited between July 2003 and January 2008.
Pre-assignment Details: Of the 166 women enrolled, 58 were found to be ineligible on clinical evaluation, 44 withdrew, and 64 were randomized.
Groups:
- Drug Therapy Alone: drug therapy alone
  Oxybutynin chloride, extended-release: Individually-titrated, extended-release oxybutynin chloride with management of side-effects.
- Drug Therapy + Behavioral Training: drug therapy + behavioral training
  Oxybutynin chloride, extended-release: Individually-titrated, extended-release oxybutynin chloride with management of side-effects.
  Behavior Training: Behavioral training consists of teaching urge suppression strategies and pelvic floor muscle training.
Period: Overall Study
Arm/Group | Drug Therapy Alone | Drug Therapy + Behavioral Training
Started | 32 | 32
Completed Therapy | 31 | 28
Completed Post-treatment Assessment | 31 | 27
Completed 6-month Follow-up | 28 | 25
Completed | 28 | 22
Not Completed | 4 | 10

BASELINE CHARACTERISTICS:
Groups:
- Arm 1: drug therapy alone
  Extended release Oxybutynin Chloride : Individually-titrated, extended release oxybutynin chloride with management of side-effects.
- Arm 2: drug therapy + behavioral training
  Extended release Oxybutynin Chloride : Individually-titrated, extended release oxybutynin chloride with management of side-effects.
  Behavior Training : Behavioral training consists of teaching urge suppression strategies and pelvic floor muscle training.
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Total
Number analyzed (Participants) | 32 | 32 | 64
Age Continuous [Mean (Standard Deviation); unit: years] | 59.3 (11.2) | 57.4 (12.6) | 58.4 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 32 | 64
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 32 | 32 | 64
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 14 | 20
  White | 26 | 18 | 44
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 32 | 32 | 64
Incontinence type [Number; unit: participants]
  Urge only | 25 | 26 | 51
  Mixed urge + stress | 7 | 5 | 12
  missing | 0 | 1 | 1
Incontinence severity [Number; unit: participant]
  Mild (less than 5 episodes/wk) | 4 | 4 | 8
  Moderate (5-10 episodes/wk) | 7 | 10 | 17
  Severe (> 10 episodes/wk) | 21 | 18 | 39

OUTCOME MEASURES:

1. Primary Outcome: Change in Incontinent Episodes Immediately Post-treatment
Description: Percent change from baseline in weekly frequency of incontinent episodes immediately post-treatment, derived from baseline and week 8 seven-day bladder diaries.
Time Frame: Baseline and immediately post-treatment - week 8
Population: Intention to treat
Measure: Mean (Standard Deviation); unit: percentage change
Groups:
- Drug Therapy Alone: Extended release Oxybutynin Chloride : Individually-titrated, extended release oxybutynin chloride with management of side-effects.
- Drug Therapy + Behavioral Training: Extended release Oxybutynin Chloride : Individually-titrated, extended release oxybutynin chloride with management of side-effects.
  Behavior Training : Behavioral training consists of teaching urge suppression strategies and pelvic floor muscle training.
Arm/Group | Drug Therapy Alone | Drug Therapy + Behavioral Training
Number analyzed (Participants) | 32 | 32
percentage change | -88.5 (24.0) | -78.3 (32.6)
Statistical Analysis 1: Comparison: Drug Therapy Alone vs Drug Therapy + Behavioral Training; The effectiveness of each intervention was calculated by comparing the weekly frequency of incontinent episodes (derived from seven-day bladder diaries) during baseline to that in the immediate post-intervention period (week 8). The primary analysis was based on intent-to-treat, in which post-treatment frequency of incontinence for non-completers was derived from the most recent week of diaries; Test type: Superiority or Other; p = .16, ANCOVA; ANCOVA, with baseline frequency of incontinent episodes as the covariate, was used to compare the treatment groups; Mean Difference (Final Values) = 10.2, 95% CI 2-sided [-5.13 to 25.54], Standard Error of Mean 7.65

2. Secondary Outcome: Change in Incontinent Episodes at 12-month Follow-up
Description: Percent change from baseline in weekly frequency of incontinent episodes at 12-months post-treatment, derived from baseline and 12-month seven-day bladder diaries
Time Frame: Baseline and 12 months post-treatment
Population: Intention to treat
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Drug Therapy Alone | Drug Therapy + Behavioral Training
Number analyzed (Participants) | 32 | 32
percent change | -82.0 (26.1) | -75.2 (33.4)
Statistical Analysis 1: Comparison: Drug Therapy Alone vs Drug Therapy + Behavioral Training; Test type: Superiority or Other; p = .37, ANCOVA; ANCOVA, with baseline frequency of incontinent episodes as the covariate, was used to compare the treatment groups; Mean Difference (Final Values) = 6.8, 95% CI 2-sided [-10.73 to 24.33], Standard Error of Mean 8.71

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Arm 1 | Arm 2
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 0/32 | 0/32

LIMITATIONS AND CAVEATS:
Secondary objectives could not be achieved because, based on a conditional power calculation, the trial was stopped early for futility.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes